CLINICAL TRIAL: NCT01935388
Title: Common Canister Protocol for Metered Dose Inhaler Administration in Mechanically Ventilated Patients
Brief Title: Common Canister Protocol for Inhaler Administration in Mechanically Ventilated Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Peggy Watts, MD, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJH CCP
Record Dates: First submitted 2013-07-31; First posted 2013-09-05 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-10

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Mechanical ventilation; chronic obstructive pulmonary disease; asthma; common canister; MDI; ventilator associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Common canister (Experimental): Use of a single MDI (instead of assigning each patient an individual MDI) for multiple mechanically ventilated patients. Inhalers will undergo a stringent cleaning protocol between administrations and storage.
  Interventions: Other: Common canister
- Control (No Intervention): Each patient will be assigned an individual inhaler as per standard of care practice.

INTERVENTIONS:
Other: Common canister — Drug administration via a shared canister with a standardized cleaning protocol.
  Arms: Common canister

SUMMARY:
Many hospitals employ a common canister inhaler protocol in patients that do not require mechanical ventilator support. Common canister refers to a single inhaler paired with standardized cleaning methods for use on more than one patient. Small reports suggest that this method does not pose an increased infectious risk and is associated with significant cost savings.

Common canister protocols offer a solution to the discordance between inhaler sizes and average inpatient use of the drugs. Metered dose inhaler canisters are contain enough drug for several days to weeks of daily use. However, the average length of stay for most inpatients is only several days. Therefore, most inpatients do not use all of the canister contents, an unused resource that is potentially wasted.

The common canister approach has not been previously described in mechanically ventilated patients (people requiring intensive care unit admission on breathing machines). This study aims to assess the safety of common canister utilization by assessment and comparison of infection rates in the study and control group.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated patients prescribed bronchodilator therapy in a medical intensive care unit

Exclusion Criteria:

* lung transplant
* neutropenic
* contact isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Ventilator-associated pneumonia (VAP) | 48 hours after intubation
  Pneumonia that developed in association with mechanical ventilation

SECONDARY OUTCOMES:
Inhaler drug cost | During period of mechanical ventilation, which varies depending on patient's severity of illness and reason for intubation; on average may range from 3-5 days.
  Inhaler charges accrued during mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Marin Kollef, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Gowan M, Bushwitz J, Watts P, Silver PC, Jackson M, Hampton N, Kollef MH. Use of a Shared Canister Protocol for the Delivery of Metered-Dose Inhalers in Mechanically Ventilated Subjects. Respir Care. 2016 Oct;61(10):1285-92. doi: 10.4187/respcare.04550. Epub 2016 May 3. PMID 27143787